CLINICAL TRIAL: NCT06301802
Title: Urological Outcomes of Proactive Management of Children With Myelomeningocele
Brief Title: Outcomes of Proactive Management of Children With Myelomeningocele
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Mahmoud Abdellah, assistant lecturer, Assiut University
Other Study IDs: myelomeningocele management
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Urologic Diseases
Keywords: myelomeningocele
MeSH Terms: conditions — Urologic Diseases; Meningomyelocele | interventions — Cholinergic Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CIC — clean intermittent catheterization
Drug: Anticholinergic — antimuscarinic once daily

SUMMARY:
Spina bifida birth prevalence in Africa is 0.13%. Myelomeningocele (MMC) represents the most frequent and most severe cause of NB in children. Treatment of neuropathic bladder secondary to spina bifida is an ongoing challenge. Damage of the renal parenchyma in children with NB is preventable given adequate evaluation, follow-up and proactive management. Proactive management was defined as use of clean intermittent catheterization (CIC), and/or anticholinergics at presentation, or based on initial high-risk urodynamic findings by 1 year of age. The proactive approach to treat SB (CIC and pharmacotherapy) has contributed to decreasing chronic kidney disease (CKD). Myelomeningocele is considered a complex congenital disease. Hence, a multidisciplinary team is the best choice for management of spina bifida, involving neurosurgeons, orthopedic surgeons, urologists, physical medicine and rehabilitation specialists and pediatricians. Currently, children with spina bifida in Egypt must visit multiple different locations to access the complex care they need. Here, we review our experience with patients with spina bifida who will be followed with this team with an emphasis on patients' upper urinary tract protection and decreasing urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* all patients with myelomeningocele attending Assiut university urology hospital.

Exclusion Criteria:

* Associated other urological congenital anomalies (e.g., PUV or bladder exstrophy)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients with myelomeningocele attending Assiut university urology hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
upper tract affection | 2 years
  percentage of patients developing upper tract dilatation and febrile UTI

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Elderwy, prof, Study Chair — prof of urology assiut university
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Oumer M, Taye M, Aragie H, Tazebew A. Prevalence of Spina Bifida among Newborns in Africa: A Systematic Review and Meta-Analysis. Scientifica (Cairo). 2020 Oct 6;2020:4273510. doi: 10.1155/2020/4273510. eCollection 2020. PMID 33083093
- [Background] Sager C, Barroso U Jr, Bastos JM Netto, Retamal G, Ormaechea E. Management of neurogenic bladder dysfunction in children update and recommendations on medical treatment. Int Braz J Urol. 2022 Jan-Feb;48(1):31-51. doi: 10.1590/S1677-5538.IBJU.2020.0989. PMID 33861059
- [Background] Elagami H, Abbas TO, Evans K, Murphy F. Management of neuropathic bladder secondary to spina bifida: Twenty years' experience with a conservative approach. Front Pediatr. 2022 Jul 29;10:913078. doi: 10.3389/fped.2022.913078. eCollection 2022. PMID 35967567
- [Background] Cui X, Zhao Z, Zhang T, Guo W, Guo W, Zheng J, Zhang J, Dong C, Na R, Zheng L, Li W, Liu Z, Ma J, Wang J, He S, Xu Y, Si P, Shen Y, Cai C. A systematic review and meta-analysis of children with coronavirus disease 2019 (COVID-19). J Med Virol. 2021 Feb;93(2):1057-1069. doi: 10.1002/jmv.26398. Epub 2020 Sep 28. PMID 32761898